CLINICAL TRIAL: NCT04042181
Title: A Randomised, Double-blinded, Parallel, Placebo-controlled Study to Evaluate the Effects of 12-weeks Supplementation of a Probiotic, Bif. Longum, on BMI and Anthropometric Outcomes in Overweight/Obese Adults.
Brief Title: The Effects of Supplementation of a Probiotic, B. Longum, on BMI and Anthropometric Outcomes in Overweight/Obese Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Cork (Other)
Collaborators: Atlantia Food Clinical Trials (Industry); CREMO SA (Unknown)
Responsible Party: Principal Investigator, Prof Ted Dinan, Professor and Chair of Psychiatry, PI APC Microbiome Ireland, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-088
Record Dates: First submitted 2018-11-20; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Bifidobacterium longum (Active Comparator)
  Interventions: Dietary Supplement: Bifidobacterium longum

INTERVENTIONS:
Dietary Supplement: Placebo — standard food grade excipients
  Arms: Placebo
Dietary Supplement: Bifidobacterium longum — Target dose of 1x10^10 CFU/day, plus standard food grade excipients
  Arms: Bifidobacterium longum

SUMMARY:
Obesity levels worldwide have tripled since the mid 1070's. Obesity and its co-morbidities, metabolic syndrome, type II diabetes, and cardiovascular disease, are serious widespread health concerns which urgently need to be addressed. G protein-coupled receptors (GPCRs), such as the ghrelin receptor (GHS-R1a), are well known for their key role in the homeostatic control of food intake and energy balance. Ghrelin is the major hunger hormone in the body and ghrelin-receptor antagonists have been advanced as potential anti-obesity agents. This receptor is therefore an ideal target for orally delivered probiotic-derived bioactives with excellent bioavailability. Bacterial strains with the ability to modulate these receptors may have high potential as probiotics with the ability to induce appetite modulation effects.

Due to promising pre-clinical results, the investigators aim to trial a Bif Longum probiotic, which can target these receptors, in an obese human population. We hypothesise that the probiotic will positively alter the gut-brain axis, improving control of hunger and satiety signalling adults with high BMI, leading to decreased BMI and waist-hip ratio scores. Furthermore, the investigators expect that the mechanism through which the probiotic is having a positive impact can be determined via investigation of the microbiota composition, gut hormone levels and circulating immune profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Give written informed consent;
2. Be between 18 and 65 years of age;
3. Has a BMI of between 28.0 - 34.9 Kg/m2;
4. Have a waist-hip ratio of ≥0.88 for males and ≥0.83 for females
5. Is in general good health, as determined by the investigator;
6. Willing to consume the investigational product daily for the duration of the study.

Exclusion Criteria:

1. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
   * child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 7. The subject must also agree to one of the following methods of contraception: i. Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or, ii. has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or, iii. sexual partner(s) is/are exclusively female or, iv. Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication).

     v. Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or, vi. Use of any intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study.
2. Subject regularly takes probiotics;
3. Subject is hypersensitive to any of the components of the test product;
4. Subject is severely immuno-compromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or underwent chemotherapy or radiotherapy within the last year);
5. Subject has Type 1 or Type 2 Diabetes Mellitus;
6. Subject has a history of bariatric surgery;
7. Subject has taken anti-obesity medication in the 12-weeks prior to randomisation
8. Subject is actively or has recently (3 months prior to randomisation) participated in a weight loss program or weight change of 3 kg during the past 3 months
9. Subject has a life-threatening illness
10. Subject is on a Metaformin, anti-psychotic drugs or any medication that the investigator determines could impact the results of the study; subject has commenced use within 3-months of randomization anti-hypertensive drugs, anti-depressive drugs, statin or any other medication that the investigator determines could impact the results of the study.
11. Subject has a history of co-existing gastrointestinal, and/or gynecological, and/or urologic pathology (e.g. colon cancer, colitis, Crohn's Disease, Celiac, Endometriosis, prostate cancer) or lactose intolerance;
12. Subject has a history of drug and/or alcohol abuse at the time of enrolment
13. Subject is currently, or planning, to participate in another study during the study period
14. Subject has a history of non-compliance
15. Subjects who have been on antibiotics in the 12-weeks prior to randomisation
16. Subject consumes vitamin D supplements >5000 IU/d

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMI measurement | From week-zero to week 12
  Significant change from week-zero to week-12 between active and placebo groups in percentage increase/decrease BMI

SECONDARY OUTCOMES:
Change in Waist:Hip ratio | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in waist:hip ratio
Change in serum insulin concentration | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in serum insulin concentration
Change in plasma HbA1c concentration | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in plasma HbA1c concentration
Change in plasma glucose concentration | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in plasma glucose concentration
Change in peripheral blood total cholesterol | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in peripheral blood total cholesterol
Change in peripheral blood triglycerides | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in peripheral blood total triglycerides
Change in peripheral blood HDL | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in peripheral blood HDL
Change in peripheral blood direct LDL | Significant changes from week-zero to week 6 and 12
  Significant changes from week-zero to week 6 and 12 between active and placebo groups in peripheral blood direct LDL

CONTACTS AND LOCATIONS:
Overall Officials: Ted Dinan, Principal Investigator — University College Cork
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided